CLINICAL TRIAL: NCT02888886
Title: Role of Systemic Inflammation in Increase of Cardio-vascular Risk in Chronic Obstructive Pulmonary Disease
Acronym: BPCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2006-A00053-48
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: systemic inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tobacco Products; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COPD (Experimental)
  Interventions: Other: Questionnaires about food habits and tobacco; Other: Spirometry; Other: Carotid echography; Other: Blood sample

INTERVENTIONS:
Other: Questionnaires about food habits and tobacco
Other: Spirometry
Other: Carotid echography
Other: Blood sample — for genetic polymorphism analysis, CRP, homocysteine and cytokine tests, glycemia and dyslipidemia analyses

SUMMARY:
The purpose is to study the correlation between systemic inflammation (serum levels of CRP, IL-1beta, IL-6 and TNF-alpha) or hyperhomocysteinemia and the increase of mortality, in a representative cohort of patients with chronic obstructive pulmonary disease (COPD).

Secondary purposes are:

1. To confirm the increase of cardiovascular mortality and the importance of cardiovascular morbidity in patients with COPD,
2. To establish the role of various genetic polymorphisms in the correlation between systemic inflammation and cardiovascular disorders observed in COPD,
3. To search for acceleration of aging of cardiovascular system evaluated with carotid intima-media thickness when systemic inflammation markers are increased,
4. To study the correlation between COPD risk factors (tobacco and other food factors), change of respiratory functional data and cardiovascular morbi-mortality. In this study cardiovascular morbi-mortality is defined by following disorders: ischemic cardiopathy, left-sided heart failure, cardiac arrhythmia and cerebrovascular accident. Diagnosis is confirmed with standard techniques and independently of this study. Results of clinical examination, ECG, echocardiography and /or brain scanner will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Actual or past active smoking of at least 20 packets/year
* FEV1/FVC < 70%

Exclusion Criteria:

* Co-morbidity except essential arterial hypertension controlled by treatment, stable coronary disease, type 2 diabetes and/or degenerative arthropathy (non-inflammatory rheumatic disorder)
* Acute disorder during 8 weeks before inclusion, especially COPD worsening
* Long-term corticosteroid or non-steroid anti-inflammatory treatment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2007-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Mortality | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ari CHAOUAT, Pr, Principal Investigator — Service des Maladies Respiratoires et Réanimation Respiratoire- Hôpital de Brabois- CHRU de Nancy

IPD SHARING:
Plan to Share IPD: No